CLINICAL TRIAL: NCT02563197
Title: An Open, Multi-center Study to Measure Inhaled Flow Rates Generated by Non-CF Bronchiectasis Patients for the T-326 Inhaler
Brief Title: Inhalation Flow Rate-study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17607; CIV-15-07-013749 (Other: EUDAMED No)
Record Dates: First submitted 2015-09-18; First posted 2015-09-30 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Bronchiectasis
Keywords: Device study; Peak inspiratory flow rate; Non-cystic fibrosis bronchiectasis; T-326 Inhaler
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T-326 (Experimental): Non Cystic fibrosis bronchiectasis patients will be enrolled for determination of peak inspiratory flow.
  Interventions: Device: T-326 Inhaler

INTERVENTIONS:
Device: T-326 Inhaler — No drug dosing,three test inhalations through the inhaler device filled with an empty capsule.

SUMMARY:
Study should show feasibility of the device for drug delivery into the lung independently of the severity of impaired lung function.

DETAILED DESCRIPTION:
The aim of the study is to measure inspiratory profiles of patients with non-Cystic fibrosis bronchiectasis using the breath activated T-326 Inhaler.

The following parameters will be derived from the inspiratory profiles:

* Peak Inspiratory Flow (PIF, in L/min)
* Inspiratory Volume (V, in L)
* Inspiratory Time (t, in s).

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of non-cystic fibrosis bronchiectasis, confirmed and documented by high resolution computed tomography (HRCT) or magnetic resonance tomography (MRT)
* Ability to reproducibly perform spirometry according to American Thoracic Society/European Respiratory Society criteria
* Clinically stable in the opinion of the investigator at the time of the study visit.
* Male and female patients ≥ 18 years of age.

Exclusion Criteria:

* Pulmonary exacerbation (as judged by the investigator, based on the clinical condition of the subject and taking into account e.g., febrile infection of the lung, relevant decrease in Forced expiratory volume in the first second (FEV1) value, increased sputum production, sputum purulence, recent hospitalization) at study visit or within the preceding six (6) weeks.
* History of lung transplant.
* Recent significant hemoptysis (≥ 300 mL or requiring blood transfusion) in the preceding six (6) weeks before screening.
* Established diagnosis of bronchial asthma.
* Established diagnosis of cystic fibrosis.
* Proof of any relevant medical finding or disease in the last three (3) months which might interfere with participation in the study or patient safety (e.g. pneumothorax, uncontrolled hypertension, uncontrolled cardiac arrhythmia, myocardial infarction, cerebral vascular accident).
* A relevant disease that is considered to interfere with the study results is any disease that, except for the impairment of lung function, interferes with the patient's ability to inhale from the device. For example, COPD per se is usually not considered as a reason for patient exclusion, unless coughing or obliteration of the upper airways with sputum interferes with the patient's ability to inhale from the device.
* Relevant surgical history in the last 3 months (e.g., but not limited to abdominal, thoracic, ocular or brain surgery).
* History or evidence of lung resection, thoracotomy, known aneurysm and severe scoliosis.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Peak inspiratory flow (L/min) | Visit 2 (1-14 days after screening visit 1)

SECONDARY OUTCOMES:
Inspiratory volumes (V in L) | Visit 2 (1-14 days after screening visit 1)
Inspiratory time (t in s) | Visit 2 (1-14 days after screening visit 1)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Germany (7):
  - Gauting, Bavaria
  - Landsberg am Lech, Bavaria
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Neu-Isenburg, Hesse
  - Hanover, Lower Saxony
  - Großhansdorf

REFERENCES:
- [Derived] Stass H, Nagelschmitz J, Kappeler D, Sommerer K, Patzlaff A, Weimann B. Ciprofloxacin Dry Powder for Inhalation: Inspiratory Flow in Patients with Non-cystic Fibrosis Bronchiectasis. J Aerosol Med Pulm Drug Deliv. 2019 Jun;32(3):156-163. doi: 10.1089/jamp.2018.1464. Epub 2019 Mar 8. PMID 30848695